CLINICAL TRIAL: NCT05351580
Title: DiSCERN: Advanced PD Therapy Candidacy and Evaluation System - Advanced PD Data Collection
Brief Title: DiSCERN: Advanced PD Therapy Candidacy and Evaluation System
Acronym: DiSCERN
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of Cincinnati (Other); The Cleveland Clinic (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Ohio State University (Other)
Responsible Party: Principal Investigator, Dustin Heldman, Principal Investigator, Great Lakes NeuroTechnologies Inc.
Other Study IDs: 5R44MD013767-03 (NIH); 5R44MD013767-03 (NIH)
Record Dates: First submitted 2022-04-15; First posted 2022-04-28 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Dyskinesia; Parkinson's Disease; Deep brain stimulation; Wearable
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Advanced Parkinson's disease patients who receive advance therapy during the study: All participants will have advanced Parkinson's disease and undergo smart watch monitoring. Participants in this cohort will be those who receive advance therapy during the study.
  Interventions: Device: DiSCERN
- Advanced Parkinson's disease patients who do not receive advance therapy during the study: All participants will have advanced Parkinson's disease and undergo smart watch monitoring. Participants in this cohort will be those who do not receive advance therapy during the study.
  Interventions: Device: DiSCERN

INTERVENTIONS:
Device: DiSCERN — Smart watch Monitoring

SUMMARY:
To collect data to develop models that identify when patients with advanced Parkinson's disease (PD) are not responding well to their current therapy and may be ready to consider advanced therapy and when patients receiving advanced therapy are not responding well and need a therapy adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Diagnosed with Parkinson's disease
* Current levodopa use
* Hoehn and Yahr scale II-III
* Ambulatory and capable of using the DiSCERN smartphone system
* Able to understand and follow instructions regarding using the device
* Half of participants (10 per site) identified as candidates for deep brain stimulation or drug pump by their treating neurologist, but before their surgeries take place.
* The remainder (10 per site) will be individuals with advanced PD as defined by having a UPDRS motor complications scores ≥ 4.

Exclusion Criteria:

* Any subject that does not meet the inclusion criteria will be excluded from this study. Subjects not capable of following the required clinical instruction for this study will be excluded. Potential subjects will be screened to ensure no cognitive impairments exist that would prohibit them from properly using the system. Exclusion criteria includes cognitive impairment as evidenced by a score less than 24 on the Montreal Cognitive Assessment (MoCA) UNLESS the subject has a caregiver able and willing to facilitate use of the DiSCERN system based on the judgement of the treating neurologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our three clinical sites will recruit a total of 60 individuals diagnosed with advanced PD who regularly take levodopa. At least half the subjects will have already been identified as candidates for DBS or LCIG, but before their surgeries take place. The remainder will be non-demented (MoCA > 24) advanced PD patients as defined by having a UPDRS motor complications scores ≥ 4. All participants must be ambulatory and capable of using the smartphone-based DiSCERN system either independently or with the help of a caregiver.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Symptom severities | Eight (8) months compared to baseline
  Symptom severities measured by smart watch

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) Part III | Eight (8) months compared to baseline
  UPDRS Part III has 33 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Each of the 33 items in the UPDRS part III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The motor score ranges from 0 to 132, where the maximum score indicates the worse condition. A negative value in change indicates improvement, whereas a positive value indicates worsening of disease.
Kinesia ONE motor assessment | Eight (8) months compared to baseline
Parkinson's Disease Questionnaire (PDQ-39) | Eight (8) months compared to baseline
  The PD Quality of Life Questionnaire-39 (PDQ-39) is a self-report questionnaire that examines health related difficulties specific to PD in eight quality of life categories within the last month. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100, with higher % indicating more health problems.
Montreal Cognitive Assessment (MoCA) | Eight (8) months compared to baseline
  The MoCA consists of 30 test items that assess visuospatial and executive functioning, naming, memory, attention, language, abstraction, delayed recall, and orientation. Each correct answer is awarded one point, which are added to create a total score. A higher score is a better outcome and indicates less cognitive impairment.
MANAGE-PD questionnaire | Eight (8) months compared to baseline
  MANAGE-PD is designed to support healthcare providers in the identification of patients with Parkinson's Disease uncontrolled on oral medications. The questionnaire consists of two sections and should be answered based on symptoms during the last month. Patients are categorized into three categories based on responses:
  Category 1: Patient may be controlled on the current treatment regimen. Category 2: Patient may not be controlled on the current treatment regimen. Category 3: Patient may not be controlled on the current treatment regimen and may benefit from device-aided therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heldman DA, Giuffrida JP, Cubo E. Wearable Sensors for Advanced Therapy Referral in Parkinson's Disease. J Parkinsons Dis. 2016 Jul 2;6(3):631-8. doi: 10.3233/JPD-160830. PMID 27392872